CLINICAL TRIAL: NCT04544865
Title: A Prospective, Single-Arm, Multi-Center Study of the ECHELON ENDOPATH(TM) Staple Line Reinforcement Device in Gastric and Lung Resection Procedures
Brief Title: Study of ECHELON ENDOPATH(TM) Staple Line Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESC_2018_03
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Gastric Procedures; Lung Resection Procedures
Keywords: Buttress, gastrectomy, gastric bypass, lung volume reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gastric and thoracic staple line reinforcement (Experimental): ECHELON ENDOPATH Staple Line Reinforcement is used during a gastric or thoracic procedure.
  Interventions: Device: Staple Line Reinforcement

INTERVENTIONS:
Device: Staple Line Reinforcement — ENDOPATH ECHELON Staple Line Reinforcement is used for reinforcement of staple lines during lung resection and bariatric surgical procedures, according to instructions for use.

SUMMARY:
This prospective, single-arm, multi-center evaluation will collect clinical data in a post-market setting. The two types of procedures studied will be gastric and thoracic. Investigators will perform each procedure using the device in compliance with their standard surgical approach and the ECHELON ENDOPATH Staple Line Reinforcement instructions for use.

DETAILED DESCRIPTION:
The primary objective of this study is to prospectively generate clinical data on device-related adverse events in a post-market setting using ECHELON ENDOPATH Staple Line Reinforcement per its instructions for use. There will be no blinding in this study. An interim analysis is planned for sample-size re-estimation.

ELIGIBILITY:
Inclusion Criteria:

* Primary procedure (gastric or lung resection) where the ECHELON SLR is planned to be used for reinforcement of staple lines per the IFU in either a or b:

  1. Gastric procedures limited to laparoscopic gastric resection, robotic laparoscopic gastric resection, partial gastrectomy, gastric wedge resection, subtotal gastrectomy, laparoscopic Roux-en-Y gastric bypass, and robotic laparoscopic gastric bypass; or
  2. Lung resection procedures that include lobectomy, segmentectomy or wedge resection, and lung volume reduction surgery, and may be video assisted thoracic surgery (VATS) or open procedures;
* Willingness to give consent and comply with all study-related evaluations and visit schedule; and
* At least 18 years of age.

Exclusion Criteria:

- Preoperative:

1. Physical or psychological condition which would impair study participation;
2. Body mass index (BMI) ≥ 46.0 kg/m2;
3. The procedure is a revision/reoperation for the same indication or same anatomical location;
4. A procedure where extended wound or organ support is required;
5. Any medical condition that the investigator deems could impact inflammatory or immune response;
6. Concurrent treatment with medications that the investigator deems could have influence on wound healing;
7. History of hypersensitivity to polyglactin (Vicryl®), Polydioxanone (PDO or PDS), or hypersensitivity to related products (cross-allergy); or
8. Enrollment in a concurrent interventional clinical study that could impact the study endpoints.

   * Intraoperative:
9. Per surgeon discretion, presence of adhesions that could lead to an increased risk of leak occurrence at a different location than the staple line.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Popoff, MD, Principal Investigator — Henry Ford Health System; David Zeltsman, MD, Principal Investigator — Long Island Jewish Medical Center; Andrew Wheeler, MD, Principal Investigator — University of Missouri-Columbia; Jon Schram, MD, Principal Investigator — Corewell Health West; Kenneth Kesler, MD, Principal Investigator — Indiana University Health; Emily Cassidy, MD, Principal Investigator — Our Lady of the Lake Hospital; Keith Gersin, MD, Principal Investigator — Wake Forest University Health Sciences; Linda Martin, MD, Principal Investigator — University of Virginia
Locations (8):
- United States (8):
  - Indiana University Health, Indianapolis, Indiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Missouri, Columbia, Missouri
  - Long Island Jewish Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who planned to have an elective gastric or lung resection surgical procedure were recruited in the study.
Pre-assignment Details: Participants were screened anytime during a period of 8 weeks prior to the date of surgery.
Groups:
- Gastric Participants: Gastric participants were treated with at least one ECHELON ENDOPATH Staple Line Reinforcement (SLR) during elective resection procedure and were followed post-operatively through discharge and at post-surgery through 70 days.
- Thoracic Participants: Thoracic participants were treated with at least one ECHELON ENDOPATH SLR during elective resection procedure and were followed post-operatively through discharge and at post-surgery through 70 days.
Period: Overall Study
Arm/Group | Gastric Participants | Thoracic Participants
Started | 109 | 131
Completed | 98 | 120
Not Completed | 11 | 11
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 11 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Participants | Thoracic Participants | Total
Number analyzed (Participants) | 109 | 131 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (11.3) | 62.8 (12.0) | 54.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 73 | 164
  Male | 18 | 58 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 99 | 122 | 221
  Unknown or Not Reported | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 85 | 108 | 193
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Specific Device-related Adverse Events (AEs) Through 70 Days Post Gastric Resection Procedures
Description: Number of participants who experienced specific device-related AEs post gastric resection procedures was reported. Specific device-related AEs were bleeding (defined as occurrence of post-surgery blood transfusion deemed related to bleeding at the staple line or return to surgery room before 70-day post-surgery follow-up visit due to bleeding deemed related to the staple line), leak (defined as occurrence of intra-surgery or post-surgery gastrointestinal leak related to the staple line as documented intra-surgery, by clinical exam, or radiographically), and stricture (defined as occurrence of stricture documented radiographically or by endoscopy along the staple line).
Time Frame: From Day 0 (day of surgery) through 70 days post-surgery
Population: The analysis set included all participants in whom the ECHELON SLR was utilized during the surgical procedure and completed the study through 70-days. Here, N' (number of participants analyzed) signifies the participants who were evaluable for this outcome measure. This outcome measure was planned to be analyzed for specified arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Gastric Participants
Number analyzed (Participants) | 104
Participants
  Bleeding | 0
  Leak | 1
  Stricture | 0

2. Primary Outcome: Number of Participants Who Experienced Specific Device-related Adverse Events Through 70 Days
Description: Number of participants who experienced specific device-related AEs post lung resection procedures was reported. Specific device related AEs were prolonged air leak (occurrence of intra-surgery or post-surgery lung leak related to the staple line as documented intra-surgery, by clinical exam, or radiographically) deemed related to the staple line (greater than post-surgery Day 7), and empyema (defined as purulent fluid collection in the pleural space documented radiographically, excluding chronic empyema).
Time Frame: From Day 0 (day of surgery) through 70 days post-surgery
Population: The analysis set included all participants in whom the ECHELON SLR was utilized during the surgical procedure and completed the study through 70-days. This outcome measure was planned to be analyzed for specified arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Participants
Number analyzed (Participants) | 131
Participants
  Prolonged air leak | 0
  Empyema | 0

3. Secondary Outcome: Number of Study Devices Replaced During Surgery
Description: Number of study devices replaced during surgery due to slipping or bunching or not properly loaded onto stapler cartridge, Other - preloaded wrong color cartridge, Other- SLR added before cartridge, Other- dropped on the ground was reported.
Time Frame: Day 0 (Intra-surgery)
Population: The analysis set included all participants in whom the ECHELON SLR is utilized during the surgical procedure.
Measure: Number; unit: Replaced study devices
Units Other Than Participants: Study devices
Arm/Group | Gastric Participants | Thoracic Participants
Number analyzed (Participants) | 109 | 131
Number analyzed (Study devices) | 637 | 598
Replaced study devices
  Slipping | 0 | 3
  Bunching | 0 | 1
  Not Loaded Properly | 7 | 3
  Other - Preloaded Wrong Color Cartridge | 1 | 0
  Other- SLR Added Before Cartridge | 1 | 0
  Other- Dropped on the Ground | 1 | 0

4. Secondary Outcome: Device Usability Evaluation by Surgeon Questionnaire: Investigator's Device Experience Feedback
Description: Investigators were asked to answer a non-validated device questionnaire related to his/her experience using the ECHELON SLR. Questionnaire included following questions "experienced less manipulation or movement compared to previous device, experienced greater confidence the device will deliver best result compared to previous device, experienced greater confidence in simplicity of set up compared to previous device, experienced less frustration with device compared to previous device, experienced less waste compared to previous device, Likely to recommend to a colleague. Each question response was ranged from 1 to 5 where 1=strongly disagree, 2=slightly disagree,3=neutral, 4=slightly agree, 5= strongly agree, where the higher response signified good experience on the device. In this outcome measure, device questionnaire responses which were provided by selected investigators after the site's first, third, and 5th procedure were reported.
Time Frame: Day 0 (Intra-surgery)
Population: The analysis set included all participants in whom the ECHELON SLR is utilized during the surgical procedure. Here, 'N' (number of participants analyzed) signifies the number of investigators who responded to device questionnaire.
Measure: Number; unit: Investigators
Arm/Group | Gastric Participants | Thoracic Participants
Number analyzed (Participants) | 12 | 18
Investigators
  Experienced less buttress manipulation and movement compared to previous buttress: Strongly disagree | 0 | 1
  Experienced less buttress manipulation and movement compared to previous buttress: Slightly disagree | 0 | 1
  Experienced less buttress manipulation and movement compared to previous buttress: Neutral | 3 | 1
  Experienced less buttress manipulation and movement compared to previous buttress: Slightly agree | 6 | 2
  Experienced less buttress manipulation and movement compared to previous buttress: Strongly agree | 3 | 13
  Greater confidence that SLR buttress deliver best outcomes compared to previous: Strongly disagree | 0 | 0
  Greater confidence that SLR buttress deliver best outcomes compared to previous:Slightly disagree | 3 | 0
  Greater confidence that SLR buttress deliver best outcomes compared to previous: Neutral | 6 | 0
  Greater confidence that SLR buttress deliver best outcomes compared to previous: Slightly agree | 2 | 2
  Greater confidence that SLR buttress deliver best outcomes compared to previous: Strongly agree | 1 | 16
  SLR setup simplifies concerns compared to previous buttress product: Strongly disagree | 0 | 0
  SLR setup simplifies concerns compared to previous buttress product: Slightly disagree | 0 | 0
  SLR setup simplifies concerns compared to previous buttress product: Neutral | 0 | 0
  SLR setup simplifies concerns compared to previous buttress product: Slightly agree | 0 | 0
  SLR setup simplifies concerns compared to previous buttress product: Strongly agree | 12 | 18
  Surgical staff experienced less frustration with SLR compared to previous buttress:Strongly disagree | 0 | 0
  Surgical staff experienced less frustration with SLR compared to previous buttress:Slightly disagree | 0 | 0
  Surgical staff experienced less frustration with SLR compared to previous buttress: Neutral | 0 | 0
  Surgical staff experienced less frustration with SLR compared to previous buttress: Slightly agree | 0 | 0
  Surgical staff experienced less frustration with SLR compared to previous buttress: Strongly agree | 12 | 18
  Foresee less waste of SLR compared to the previous buttress: Strongly disagree | 0 | 0
  Foresee less waste of SLR compared to the previous buttress: Slightly disagree | 1 | 0
  Foresee less waste of SLR compared to the previous buttress: Neutral | 1 | 2
  Foresee less waste of SLR compared to the previous buttress: Slightly agree | 4 | 2
  Foresee less waste of SLR compared to the previous buttress: Strongly agree | 6 | 14
  Likely to recommend to a colleague: Strongly disagree | 0 | 0
  Likely to recommend to a colleague: Slightly disagree | 0 | 0
  Likely to recommend to a colleague: Neutral | 0 | 0
  Likely to recommend to a colleague: Slightly agree | 5 | 2
  Likely to recommend to a colleague: Strongly agree | 7 | 16

5. Secondary Outcome: Device Usability Evaluation by Surgeon Questionnaire: Investigator's Device Satisfaction Feedback
Description: Investigators were asked to answer a non-validated device questionnaire related to his/her experience using the ECHELON SLR. Questionnaire included following questions "satisfaction of operative flow compared to previous device and satisfaction of manipulation and repositioning compared to previous device" and each question response was ranged from 1 to 5 where 1=very dissatisfied, 2=dissatisfied, 3=neither dissatisfied nor satisfied (NDNS), 4=satisfied, 5=very satisfied, where higher response signified good satisfaction with the device. In this outcome measure, device questionnaire responses which were provided by selected investigators after the site's first, third, and fifth procedure were reported.
Time Frame: Day 0 (Intra-surgery)
Population: The analysis set included all participants in whom the ECHELON SLR is utilized during the surgical procedure. Here, N' (number of participants analyzed) signifies the number of investigators who responded to device questionnaire.
Measure: Number; unit: Investigators
Arm/Group | Gastric Participants | Thoracic Participants
Number analyzed (Participants) | 12 | 18
Investigators
  Satisfaction of operative flow compared to previous device: Very dissatisfied | 0 | 0
  Satisfaction of operative flow compared to previous device: Dissatisfied | 0 | 0
  Satisfaction of operative flow compared to previous device: Neither dissatisfied nor satisfied | 0 | 0
  Satisfaction of operative flow compared to previous device: Satisfied | 3 | 2
  Satisfaction of operative flow compared to previous device: Very satisfied | 9 | 16
  Satisfaction of manipulation and repositioning compared to previous device:Very dissatisfied | 0 | 0
  Satisfaction of manipulation and repositioning compared to previous device: Dissatisfied | 0 | 0
  Satisfaction of manipulation and repositioning compared to previous device: NDNS | 0 | 0
  Satisfaction of manipulation and repositioning compared to previous device: Satisfied | 1 | 3
  Satisfaction of manipulation and repositioning compared to previous device: Very satisfied | 11 | 15

ADVERSE EVENTS:
Time Frame: From Day 0 (Day of surgery) up to end of the study (2 years 4 months)
Description: The analysis set included all participants in whom the ECHELON SLR was utilized during the surgical procedure.
Arm/Group | Gastric Participants | Thoracic Participants
All-Cause Mortality (participants affected / at risk) | 0/109 | 2/131
Serious Adverse Events (participants affected / at risk) | 8/109 | 18/131
Other Adverse Events (participants affected / at risk) | 74/109 | 116/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Participants (N=109) | Thoracic Participants (N=131)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Fistulas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Gastric Participants (N=109) | Thoracic Participants (N=131)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 66 (71)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 42 (42)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 34 (37)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 17 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 34 (39) | 12 (12)
Vomiting (Gastrointestinal disorders) | 24 (26) | 4 (4)
Constipation (Gastrointestinal disorders) | 12 (12) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 11 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 8 (8) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2)
Eructation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal fat apron (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 62 (62)
Incision site pain (Injury, poisoning and procedural complications) | 8 (9) | 5 (5)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-thoracotomy pain syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 21 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 8 (8)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 1 (1) | 1 (1)
Administration site swelling (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 8 (8)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pneumopericardium (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (2)
Thoracic cavity drainage test abnormal (Investigations) | 0 (0) | 2 (2)
Chest X-ray (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 0/109 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT04544865/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT04544865/SAP_001.pdf